CLINICAL TRIAL: NCT05055999
Title: Tumor Microenvironment Surveillance on Simultaneous Liver Metastases Extensive Stage Small Cell Lung Cancer Who Treated With Atezolizumab Plus Etoposide and Platinum Based Chemotherapy
Brief Title: Tumor Microenvironment Surveillance on Simultaneous Liver Metastases Extensive Stage Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Other Study IDs: MATCH
Record Dates: First submitted 2021-09-15; First posted 2021-09-24 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2019-04

CONDITIONS: Extensive Stage Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — FFPE: RNA-seq, WES, and Multi-immunofluorescence based IHC, Spatial transcriptomics Plasma+PBMC: Cytokine/chemokines and TCR-seq Fecal microbiota: Metabolomics and Metagenomic sequencing Fresh tissue Fresh tissue: RNA-seq? TCR? WES? Metabolomics? Single Cell Sequence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: First line EC/EP+Atezolizumab — Etoposide (100mg/㎡) Carboplatin (AUC=4) Atezolizumab(1200mg) ivgtt, every 21 day

SUMMARY:
The purpose of the trial is to detect tumor microenvironment on Extensive Stage Small Cell Lung Cancer with simultaneous liver metastases who Treated with Atezolizumab plus Etoposide and Platinum Based Chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18， Extensive Stage Small Cell Lung Cancer Confirmed by Histopathology Treated with Atezolizumab plus Etoposide and Platinum Based Chemotherapy

Exclusion Criteria:

- Patients with contraindication of chemotherapy Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Extensive Stage Small Cell Lung Cancer who Treated with Atezolizumab plus Etoposide and Platinum Based Chemotherapy
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
PFS | April 2019- July 2021
  Progression free survival
OS | April 2019- July 2021
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China